CLINICAL TRIAL: NCT03834298
Title: Non-endoscopic Tracking of Disease Activity During Dietary Interventions in Eosinophilic Esophagitis
Brief Title: Non-endoscopic Tracking of Disease Activity in Eosinophilic Esophagitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study grant not obtained; not moving forward with study at this time.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Northwestern University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-0018
Record Dates: First submitted 2019-01-04; First posted 2019-02-07 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Four Food Elimination Diet (FFED) (Experimental): There is one arm to the study. All participants meeting eligibility will be assigned to intervention / treatment with a previously defined four food elimination diet (FFED) (Aim 1). This is a longitudinal study in which outcome measures including symptoms, QOL and inflammation at baseline and at 2, 4 and 6 weeks after starting stand of care (SOC) FFED will be measured. Participants meeting eligibility for Aim 2 will have foods added back to the diet using a specified protocol.
  Interventions: Other: Four Food Elimination Diet

INTERVENTIONS:
Other: Four Food Elimination Diet — Food allergens are thought to initiate eosinophilic inflammation and dietary elimination of trigger allergens is an effective treatment for EoE. Previous work demonstrates that in both children and adult EoE patients, the food antigens including cow's milk, wheat, egg, soy, peanut/tree nut and fish/shell fish, are the most common food triggers causing esophageal inflammation. Participants will be assigned to single arm treatment / intervention with a diet restricted of the four most common food allergens, milk, soy, wheat and egg, or a four food elimination diet (FFED). With the goal to optimize diet treatment, in Aim 2, eligible participants will undergo sequential food reintroductions based on protocol.

SUMMARY:
To prospectively determine the natural history of inflammation resolution following initiation of diet treatment and to optimize the diet treatment of patients with EoE through the use of a non-endoscopic tracking device, the esophageal string test (EST).

DETAILED DESCRIPTION:
This is an adult and pediatric prospective, longitudinal study in which we will measure symptoms, QOL and inflammation at baseline and again at 2, 4 and 6 weeks after starting stand of care (SOC) four food elimination diet (FFED) (Aim 1). Newly or previously diagnosed patients with EoE with active disease who will be undergoing SOC FFED will be offered entry into the study by the PI's or their local co-investigators at each of their institutions. EoE patients who are in remission on SOC FFED from Aim 1 will be recruited to participate in this food reintroduction trial in Aim 2. Eligible subjects will undergo SOC sequential food reintroductions and during the food introduction, ESTs will be performed at 2 and 4 week intervals during a clinic visit. If inflammation is detected by the EST, this food will be eliminated from the diet for six weeks and a repeat EST will be administered at this time to assess inflammation. If inflammation has resolved based on EST results, food reintroduction will resume. If no inflammation is detected by the EST at the 4 week interval, a new food will be added. EST will be performed after each food reintroduction as outlined above. Based on known allergenic properties of these foods, the order of food reintroduction will be soy, eggs, wheat and milk.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to understand and provide informed consent
* Males and Females ≥7 years of age to 65 years of age
* Have diagnosis of EoE
* Have histologically confirmed active disease ≥15 eosinophils/hpf
* Symptomatic (have experienced symptoms within the last one months prior to enrollment).
* Female subjects of childbearing potential must have a negative pregnancy test upon study entry
* Female (and male) subjects with reproductive potential, must agree to use FDA approved methods of birth control for the duration of the study

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Secondary causes of eosinophilia
* Pregnancy
* Immunodeficiency states
* Have participated in any investigative drug study within 6 weeks prior to study entry
* Unable to complete study procedures including endoscopy
* Luminal stricture identified <13mm which would prevent passage of the EST and prevent assessment of mucosal inflammation
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease Remission as Measured by Esophageal String Test (EST) Score (EoEScore) | 6 weeks
  Disease remission will be an EoEScore <0.36, the score below which the patient has a very low probability of having an eosinophil count > 15 eos/HPF = active EoE. This decision rule is associated with a sensitivity of 0.92 and specificity of 0.28 for having active EoE.
Disease Remission as Measured by Esophageal String Test (EST) Score (EoEScore) | 2 weeks
  Disease remission will be an EoEScore <0.36, the score below which the patient has a very low probability of having an eosinophil count > 15 eos/HPF = active EoE. This decision rule is associated with a sensitivity of 0.92 and specificity of 0.28 for having active EoE. This 2 week time point will be a co-primary outcome measure.
Disease Remission as Measured by Esophageal String Test (EST) Score (EoEScore) | 4 weeks
  Disease remission will be an EoEScore <0.36, the score below which the patient has a very low probability of having an eosinophil count > 15 eos/HPF = active EoE. This decision rule is associated with a sensitivity of 0.92 and specificity of 0.28 for having active EoE. This 4 week time point will be a co-primary outcome measure.

SECONDARY OUTCOMES:
Change in Symptom Severity in Participants Age 18-65 as Measured by Eosinophilic Esophagitis Activity Index (EESAI) | Baseline and 6 weeks
  The validated symptoms severity assessment tool Eosinophilic Esophagitis Activity Index (EESAI) will be used to assess severity in participants age 18 to 65.
Change in Symptom Severity in Participants Age 7-18 as Measured by Pediatric Eosinophilic Esophagitis Symptom Severity (PEESS v 2.) | Baseline and 6 weeks
  The validated symptoms severity assessment tool Pediatric Eosinophilic Esophagitis Symptom Severity (PEESS v 2.) will be used to assess severity in participants age 7 to 18.
Time to Disease Recurrence as Measured by EST score | 4 weeks after food re-introduction
  To determine the time to disease recurrence with re-introduction of potential food allergen triggers, disease recurrence will be indicated by an EoEScore probability of > 0.53.
Time to Disease Recurrence as Measured by EST score | 2 weeks after food re-introduction
  To determine the time to disease recurrence with re-introduction of potential food allergen triggers, disease recurrence will be indicated by an EoEScore probability of > 0.53.

CONTACTS AND LOCATIONS:
Overall Officials: Calies Menard-Katcher, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No